CLINICAL TRIAL: NCT00439725
Title: Once-daily Oral Direct Factor Xa Inhibitor Rivaroxaban in the Long-term Prevention of Recurrent Symptomatic Venous Thromboembolism in Patients With Symptomatic Deep-vein Thrombosis or Pulmonary Embolism. The Einstein-Extension Study
Brief Title: Once - Daily Oral Direct Factor Xa Inhibitor Rivaroxaban In The Long-Term Prevention Of Recurrent Symptomatic Venous Thromboembolism In Patients With Symptomatic Deep-Vein Thrombosis Or Pulmonary Embolism. The Einstein-Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11899; 2006-004494-96 (EudraCT Number)
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Results first posted 2012-04-12 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental): Participants were to receive rivaroxaban 20 mg oral tablet once daily
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Placebo (Placebo Comparator): Participants were to receive matching placebo oral tablet once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Patients randomized to rivaroxaban will receive rivaroxaban 20 mg once-daily.
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Placebo — Patients allocated to placebo will receive a matching placebo tablet once daily.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, event-driven, superiority study for efficacy. Patients with confirmed symptomatic DVT (deep vein thrombosis) or PE (pulmonary embolism) who completed 6 or 12 months of treatment with rivaroxaban or VKA (vitamin K antagonist) are eligible for this trial (Einstein-Extension study).

DETAILED DESCRIPTION:
Within the US 'Johnson & Johnson Pharmaceutical Research & Development, L.L.C.' is sponsor.

The treatment period was followed by an observational period of 30 days starting the day after the last intake of study medication, regardless of the actual duration of study drug administration. Participants who did not complete the treatment period also entered the observational period. It was also possible that participants did not enter the observational period, e.g. due to withdrawal of consent or termination of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed symptomatic PE or DVT who have been treated for 6 or 12 months with VKA or rivaroxaban

Exclusion Criteria:

* Legal lower age limitations (country specific)
* Indication for VKA other than DVT and/or PE
* Patients in whom anticoagulant treatment for their index PE or DVT should be continued
* Childbearing potential without proper contraceptive measures, pregnancy or breast feeding. Proper contraceptive measures are defined as a method of contraception with a failure rate < 1 % during the course of the study (including the observational period). These methods of contraception according to the note for guidance on non-clinical safety studies for the conduct of human trials for pharmaceuticals (CPMP [Committee for Proprietary Medicinal Products]/ICH [International Conference on Harmonization]/286/95, modification) include consistent and correct use of hormone containing implants and injectables, combined oral contraceptives, hormone containing intrauterine devices, surgical sterilization, sexual abstinence and vasectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1197 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (268):
- United States (23):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Redlands, California
  - Bay Pines, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Decatur, Georgia
  - Idaho Falls, Idaho
  - Covington, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Albuquerque, New Mexico
  - Chapel Hill, North Carolina
  - Greensboro, North Carolina
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - Corsicana, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Fredericksburg, Virginia
  - Spokane, Washington
- Australia (18):
  - Garran, Australian Capital Territory
  - Gosford, New South Wales
  - Kogarah, New South Wales
  - Lismore, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Redcliffe, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Box Hill, Victoria
  - Clayton, Victoria
  - Geelong, Victoria
  - Melbourne, Victoria
  - Prahran, Victoria
  - Fremantle, Western Australia
  - Perth, Western Australia
- Austria (5):
  - Salzburg, Salzburg
  - Graz, Styria
  - Innsbruck, Tyrol
  - Vienna, Vienna
  - Feldkirch, Vorarlberg
- Belgium (12):
  - Bruxelles - Brussel
  - Duffel
  - Genk
  - Ghent
  - Hasselt
  - Leuven
  - Lier
  - Liège
  - Namur
  - Sint-Truiden
  - Yvoir
  - Zottegem
- Brazil (8):
  - Uberaba, Minas Gerais
  - Curitiba, Paraná
  - Londrina, Paraná
  - Porto Alegre, Rio Grande do Sul
  - Botucatu, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
  - Rio de Janeiro
- Canada (2):
  - Winnipeg, Manitoba
  - Toronto, Ontario
- China (7):
  - Guangzhou, Guangdong
  - Harbin, Heilongjiang
  - Wuhan, Hubei
  - Suzhou, Jiangsu
  - Shenyang, Liaoning
  - Beijing
  - Shanghai
- Czechia (7):
  - Brno
  - Karlovy Vary
  - Kladno
  - Ostrava
  - Ostrava-Poruba
  - Prague
  - Usti Nad Lebem
- Denmark (4):
  - Aarhus C
  - Brædstrup
  - Frederiksberg
  - Hellerup
- Seinäjoki, Finland
- France (31):
  - Agen
  - Amiens
  - Angers
  - Arras
  - Bordeaux
  - Brest
  - Castelnau-le-Lez
  - Clamart
  - Clermont-Ferrand
  - Colombes
  - Créteil
  - Dijon
  - Grenoble
  - Lille
  - Limoges
  - Montpellier
  - Nantes
  - Nîmes
  - Orthez
  - Paris
  - Pierre-Bénite
  - Roanne
  - Rouen
  - Saint-Etienne
  - Strasbourg
  - Toulon
  - Toulouse
  - Tours
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vernon
- Germany (29):
  - Bruchsal, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Karlsbad, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Neckargemünd, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Augsburg, Bavaria
  - München, Bavaria
  - Würzburg, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Giessen, Hesse
  - Wiesbaden, Hesse
  - Hanover, Lower Saxony
  - Rotenburg (Wümme), Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Soest, North Rhine-Westphalia
  - Witten, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Hong Kong, Hong Kong
- Hungary (8):
  - Budapest
  - Debrecen
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Nyíregyháza
  - Szentes
  - Szombathely
- India (7):
  - Kochi, Kerala
  - Vellore, Kerala
  - Mumbai, Maharashtra
  - Hyderabad
  - Kolkata
  - New Delhi
  - Pune
- Indonesia (4):
  - Bandung
  - Jakarta
  - Medan
  - Semarang
- Israel (12):
  - Haifa, Israel
  - Petah Tikva, Israel
  - Afula
  - Ashkelon
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Rehovot
  - Safed
  - Tel Aviv
- Italy (10):
  - Bologna
  - Chieti
  - Milan
  - Napoli
  - Padua
  - Palermo
  - Parma
  - Pavia
  - Piacenza
  - Venezia
- Kuala Selangor, Malaysia
- Netherlands (11):
  - 's-Hertogenbosch
  - Amsterdam
  - Arnhem
  - Dordrecht
  - Enschede
  - Groningen
  - Hoofddorp
  - Maastricht
  - Rotterdam
  - Zwijndrecht
  - Zwolle
- New Zealand (4):
  - Auckland
  - Christchurch
  - Palmerston North
  - Wellington South
- Norway (3):
  - Fredrikstad
  - Oslo
  - Rud
- Quezon City, Philippines
- Poland (11):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- Singapore, Singapore
- South Africa (7):
  - Cape Town, Cape
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Roodepoort, Gauteng
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
- South Korea (5):
  - Daegu, Daegu Gwang'yeogsi
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Seoul
  - Taegu
- Spain (8):
  - Barcelona, Barcelona
  - Terrassa, Barcelona
  - Girona, Girona
  - Alcorcón, Madrid
  - Fuenlabrada, Madrid
  - Madrid, Madrid
  - Pamplona, Pamplona
  - Xàtiva, Valencia
- Sweden (5):
  - Borås
  - Gothenburg
  - Jönköping
  - Sundsvall
  - Västervik
- Switzerland (7):
  - Bruderholz, Basel-Landschaft
  - Zurich, Canton of Zurich
  - Genéve 14, Genève 14
  - Chur, Kanton Graubünden
  - Brig, Valais
  - Lucerne
  - Lugano
- Taiwan (4):
  - Kaohsiung City
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok, Bangkok
  - Pathumwan, Bangkok, Thailand
  - Bangkok
- United Kingdom (8):
  - Plymouth, Devon
  - Chelmsford, Essex
  - Romford, Essex
  - Isleworth, London
  - London, London
  - Edinburgh, Lothian
  - Liverpool, Merseyside
  - London

REFERENCES:
- [Result] Cohen AT, Dobromirski M. The use of rivaroxaban for short- and long-term treatment of venous thromboembolism. Thromb Haemost. 2012 Jun;107(6):1035-43. doi: 10.1160/TH11-12-0859. Epub 2012 Feb 28. PMID 22371186
- [Result] EINSTEIN Investigators; Bauersachs R, Berkowitz SD, Brenner B, Buller HR, Decousus H, Gallus AS, Lensing AW, Misselwitz F, Prins MH, Raskob GE, Segers A, Verhamme P, Wells P, Agnelli G, Bounameaux H, Cohen A, Davidson BL, Piovella F, Schellong S. Oral rivaroxaban for symptomatic venous thromboembolism. N Engl J Med. 2010 Dec 23;363(26):2499-510. doi: 10.1056/NEJMoa1007903. Epub 2010 Dec 3. PMID 21128814
- [Derived] Dobesh PP, Volkl AA, Pap AF, Damaraju CV, Levitan B, Yuan Z, Amin AN. Benefit-Risk Assessment of Rivaroxaban in Older Patients With Nonvalvular Atrial Fibrillation or Venous Thromboembolism. Drugs Aging. 2025 May;42(5):469-484. doi: 10.1007/s40266-025-01192-7. Epub 2025 Mar 31. PMID 40163217
- [Derived] Yamada N, Fu W, Shi Z, Park KH, Kim HS, Dai X, Lensing AW, Pap AF, Kohno T, Tajima T, Watakabe T, Mitsumori T. Risk of recurrent venous thromboembolism and major bleeding according to risk factor profiles in Asian patients: a subgroup analysis EINSTEIN-Extension and EINSTEIN-CHOICE. Thromb J. 2024 Jun 6;22(1):48. doi: 10.1186/s12959-024-00609-4. PMID 38844941
- [Derived] Wells PS, Prins MH, Levitan B, Beyer-Westendorf J, Brighton TA, Bounameaux H, Cohen AT, Davidson BL, Prandoni P, Raskob GE, Yuan Z, Katz EG, Gebel M, Lensing AWA. Long-term Anticoagulation With Rivaroxaban for Preventing Recurrent VTE: A Benefit-Risk Analysis of EINSTEIN-Extension. Chest. 2016 Nov;150(5):1059-1068. doi: 10.1016/j.chest.2016.05.023. Epub 2016 Jun 1. PMID 27262225
- [Derived] Wells PS, Gebel M, Prins MH, Davidson BL, Lensing AW. Influence of statin use on the incidence of recurrent venous thromboembolism and major bleeding in patients receiving rivaroxaban or standard anticoagulant therapy. Thromb J. 2014 Nov 26;12:26. doi: 10.1186/1477-9560-12-26. eCollection 2014. PMID 25698905
- See also: Click here to find the definition for Deep Vein Thrombosis [DVT]. — http://www.nhlbi.nih.gov/health/health-topics/topics/dvt/
- See also: Click here to find the definition for Pulmonary Embolism [PE]. — http://www.nhlbi.nih.gov/health/health-topics/topics/pe/
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with confirmed symptomatic deep vein thrombosis or pulmonary embolism, who either had been treated for 6 or 12 months with warfarin or acenocoumarol or rivaroxaban in study NCT00440193, or who had been treated for 6 to 14 months with warfarin or acenocoumarol outside study NCT00440193, were recruited at specialized study sites.
Pre-assignment Details: Out of 1200 participants screened, 3 failed screening (2 due to withdrawal of consent and 1 due to a protocol violation), and 1197 participants were randomized (602 to rivaroxaban and 595 to placebo).
Period: Treatment Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Started | 602 | 595
Participants Received Treatment | 598 (Safety population) | 590 (Safety population)
Completed | 366 | 349
Not Completed | 236 | 246
Not completed — Withdrawal by Subject | 22 | 19
Not completed — Study terminated by sponsor | 156 | 148
Not completed — Site closed by investigator | 1 | 2
Not completed — Adverse Event | 39 | 18
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Clinical endpoint reached | 6 | 50
Not completed — Technical problems | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Participant convenience | 1 | 0
Not completed — Protocol driven decision point | 1 | 1
Not completed — Death | 1 | 1
Not completed — Participant did not receive treatment | 4 | 4
Period: Observational Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Started | 577 (All participants who took any study medication and entered the observational period.) | 560 (All participants who took any study medication and entered the observational period.)
Completed | 569 | 553
Not Completed | 8 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 2
Not completed — Study termination by sponsor | 1 | 1
Not completed — Clinical endpoint reached | 3 | 1
Not completed — Technical problems | 1 | 0
Not completed — Participant convenience | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo | Total
Number analyzed (Participants) | 602 | 594 | 1196
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of participants analyzed for Baseline is intention-to-treat (ITT) population.
  years | 58.2 (15.6) | 58.4 (16.0) | 58.3 (15.8)
Age, Customized [Number; unit: participants] — Number of participants analyzed for Baseline is intention-to-treat (ITT) population.
  participants
    18 - 40 years | 87 | 94 | 181
    >40 - <65 years | 273 | 280 | 553
    65 - 75 years | 153 | 121 | 274
    >75 years | 89 | 99 | 188
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants analyzed for Baseline is intention-to-treat (ITT) population.
  Participants
    Female | 248 | 255 | 503
    Male | 354 | 339 | 693

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]) Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for fatal PE) or unexplained death for which DVT/PE could not be ruled out (for fatal PE), and/or case summaries. For definition of DVT/PE, kindly refer to the link in the Protocol section.
Time Frame: 6- or 12-month study treatment period
Population: The intention-to-treat (ITT) population consisted of all randomized participants with valid informed consent. Participants were analyzed according to the treatment assigned at randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 1.3 | 7.1
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Placebo; The rivaroxaban to comparator hazard ratio was computed with a 95% CI (confidence interval) (two-sided testing); Test type: Superiority or Other; p < 0.0001, Regression, Cox — 1st test in a hierarchy, a p-value of less than 0.05 would be considered significant; Stratified by intended treatment duration, adjusted for pre-treatment; Hazard Ratio (HR) = 0.185, 95% CI [0.087 to 0.393], Standard Error of Mean 0.3858

2. Secondary Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause Mortality Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), or lung scintigraphy (for PE), and/or case summaries.
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 1.3 | 7.2
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Placebo; The rivaroxaban to comparator hazard ratio was computed with a 95% CI (two-sided testing); Test type: Superiority or Other; p < 0.0001, Regression, Cox — 2nd test in a hierarchy, a p-value of less than 0.05 would be considered significant. If the 1st test in hierarchy was significant; Stratified by intended treatment duration, adjusted for pre-treatment; Hazard Ratio (HR) = 0.180, 95% CI [0.085 to 0.383], Standard Error of Mean 0.3850

3. Secondary Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE, All Cause Mortality, Strokes and Myocardial Infarctions Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 1.5 | 7.4
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Placebo; The rivaroxaban to comparator hazard ratio was computed with a 95% CI (two-sided testing); Test type: Superiority or Other; p < 0.0001, Regression, Cox — 3rd test in a hierarchy, a p-value of less than 0.05 would be considered significant. If the previous tests in hierarchy were significant; Stratified by intended treatment duration, adjusted for pre-treatment; Hazard Ratio (HR) = 0.198, 95% CI [0.096 to 0.405], Standard Error of Mean 0.3659

4. Secondary Outcome: Percentage of Participants With Net Clinical Benefit as Composite of Recurrent DVT or Non-fatal or Fatal PE and Major Bleeding Events Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound, venography, spiral computed tomography scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of ≥2 units, occurring in a critical site or contributing to death.
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 2.0 | 7.1
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Placebo; The rivaroxaban to comparator hazard ratio was computed with a 95% CI (two-sided testing); Test type: Superiority or Other; p < 0.0001, Regression, Cox — 4th test in a hierarchy, a p-value of less than 0.05 would be considered significant. If the previous tests in hierarchy were significant; Stratified by intended treatment duration, adjusted for pre-treatment; Hazard Ratio (HR) = 0.278, 95% CI [0.146 to 0.528], Standard Error of Mean 0.3274

5. Secondary Outcome: Percentage of Participants With Recurrent VTE (PE or DVT) Until the Intended End of Study Treatment
Description: as for outcome 3
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 1.2 | 7.1

6. Secondary Outcome: Percentage of Participants With Recurrent DVT Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound, venography, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 0.8 | 5.2

7. Secondary Outcome: Percentage of Participants With Major Bleeding
Description: All events were adjudicated and confirmed by a central independent adjudication committee (CIAC) blinded to treatment. Major bleeding event was overt bleeding associated with a 2 g/dL or greater fall in hemoglobin, leading to a transfusion of 2 or more units of packed red blood cells or whole blood, occurring in a critical site or contributing to death. Treatment-emergent [after intake of first tablet of study medication as randomized but not more than 2 days after stop of study medication (referred to as time window: 2 days)] events and all events post randomization were reported.
Time Frame: 6- or 12-month study treatment period
Population: The valid-for-safety analysis population consisted of all participants who were randomized with valid informed consent and received at least one dose of study treatment. For this population, participants were analyzed according to the treatment they received.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 598 | 590
Percentage of participants
  Treatment-emergent (time window: 2 days) | 0.7 | 0.0
  All post-randomization | 0.7 | 0.2
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Placebo; The rivaroxaban to comparator hazard ratio was computed with a 95% CI (two-sided testing), comparison was done for the treatment emergent (within two days after end of treatment) bleeding events; Test type: Superiority or Other; p = 0.1121, Log Rank — No adjustment for multiple comparison

8. Secondary Outcome: Percentage of Participants With Clinically Relevant Bleeding
Description: All events adjudicated/confirmed by CIAC blinded to treatment. Clinically relevant bleeding included major bleeding (definition: see outcome 7) and non-major bleeding associated with medical intervention, unscheduled physician contact, (temporary) cessation of study treatment, discomfort for the participants such as pain, or impairment of daily life activities. Treatment-emergent events (after intake of 1st study medication tablet as randomized up to 2 days after stop of study medication ['time window: 2 days']) and all events post randomization were reported
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 598 | 590
Percentage of participants
  Treatment-emergent (time window: 2 days) | 6.0 | 1.2
  All post-randomization | 6.0 | 1.9
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Cox — No adjustment for multiple comparison, a p-value of less than 0.05 would be considered significant; Stratified by intended treatment duration, adjusted for pre-treatment done for treatment-emergent (time window: 2 days); Hazard Ratio (HR) = 5.185, 95% CI [2.307 to 11.652], Standard Error of Mean 0.4131

9. Secondary Outcome: Percentage of Participants With All Death
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either autopsy, results/films/images of confirmatory testing, and/or case summaries. Treatment-emergent events and all events post randomization were reported. Treatment-emergent: after intake of first tablet of study medication as randomized but not more than 2 days after stop of study medication (referred to as time window: 2 days)
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 598 | 590
Percentage of participants
  Treatment-emergent (time window: 2 days) | 0.2 | 0.2
  All post-randomization | 0.2 | 0.3

10. Secondary Outcome: Percentage of Participants With Other Vascular Events
Description: All pre-defined vascular events (acute coronary syndromes, ischemic stroke, transient ischemic attack, non-central nervous system systemic embolism and vascular death) were adjudicated/confirmed by a central independent adjudication committee blinded to treatment, based on results/films/images of confirmatory testing, and/or case summaries. On treatment events and all events post randomization were reported. On treatment: after intake of first tablet of study medication as randomized but not more than 1 day after stop of study medication (referred to as time window: 1 day)
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 598 | 590
Percentage of participants
  On treatment (time window: 1 day) | 0.5 | 0.7
  All post-randomization | 0.8 | 0.7

11. Other Pre Specified Outcome: Percentage of Participants With Death (PE) Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either autopsy, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 0.0 | 0.2

12. Other Pre Specified Outcome: Percentage of Participants With Death (PE Cannot be Excluded) Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 0.2 | 0.0

13. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Recurrent PE Until the Intended End of Study Treatment
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either spiral computed tomography (CT) scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 6- or 12-month study treatment period
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 602 | 594
Percentage of participants | 0.3 | 2.2

14. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]) During Observational Period
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for fatal PE) or unexplained death for which DVT/PE could not be ruled out (for fatal PE), results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 30 days observational period after last intake of study medication
Population: Intention-to-treat (ITT) population entering observational period. Participants were analyzed according to the treatment assigned at randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 577 | 559
Percentage of participants | 1.2 | 0.9

15. Other Pre Specified Outcome: Percentage of Participants With Symptomatic Recurrent PE During Observational Period
Description: as for outcome 13
Time Frame: 30 days observational period after last intake of study medication
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 577 | 559
Percentage of participants | 0.3 | 0.2

16. Other Pre Specified Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause Mortality During Observational Period
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound (for DVT), venography (for DVT), spiral computed tomography (CT) scanning (for PE), pulmonary angiography (for PE), ventilation/perfusion lung scan (for PE), lung scintigraphy (for PE), autopsy (for deaths), results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 30 days observational period after last intake of study medication
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 577 | 559
Percentage of participants | 1.2 | 1.1

17. Other Pre Specified Outcome: Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE, All Cause Mortality, Strokes and Myocardial Infarctions During Observational Period
Description: as for outcome 14
Time Frame: 30 days observational period after last intake of study medication
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 577 | 559
Percentage of participants | 1.4 | 1.1

18. Other Pre Specified Outcome: Percentage of Participants With Net Clinical Benefit as Composite of Recurrent DVT or Non-fatal or Fatal PE and Major Bleeding Events During Observational Period
Description: Events were adjudicated/confirmed by a central independent adjudication committee blinded to treatment, based on either compression ultrasound, venography, spiral CT scanning, pulmonary angiography, ventilation/perfusion lung scan, lung scintigraphy, autopsy or unexplained death for which DVT/PE could not be ruled out, results/films/images of confirmatory testing, and/or case summaries. Major bleeding was overt bleeding associated with 2 g/dL or greater fall in hemoglobin, leading to a transfusion of 2 or more units, occurring in a critical site or contributing to death.
Time Frame: 30 days observational period after last intake of study medication
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 577 | 559
Percentage of participants | 1.2 | 0.9

19. Other Pre Specified Outcome: Percentage of Participants With Recurrent VTE (PE or DVT) During Observational Period
Description: as for outcome 3
Time Frame: 30 days observational period after last intake of study medication
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 577 | 559
Percentage of participants | 1.2 | 0.9

20. Other Pre Specified Outcome: Percentage of Participants With Recurrent DVT During Observational Period
Description: All events were adjudicated and confirmed by a central independent adjudication committee blinded to treatment. Events were assessed based on either compression ultrasound or venography, results/films/images of confirmatory testing, and/or case summaries.
Time Frame: 30 days observational period after last intake of study medication
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Number analyzed (Participants) | 577 | 559
Percentage of participants | 0.9 | 0.7

ADVERSE EVENTS:
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Placebo
Serious Adverse Events (participants affected / at risk) | 59/598 | 52/590
Other Adverse Events (participants affected / at risk) | 63/598 | 65/590
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=598) | Placebo (N=590)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 4
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Antiphospholipid syndrome (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Intestinal gangrene (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Postoperative abscess (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Anal fistula excision (Surgical and medical procedures) | 0 | 1
Appendicectomy (Surgical and medical procedures) | 1 | 0
Bladder calculus removal (Surgical and medical procedures) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=598) | Placebo (N=590)
Nasopharyngitis (Infections and infestations) | 33 | 32
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less